CLINICAL TRIAL: NCT04529421
Title: Relationship Between In-person Instruction and COVID-19 Incidence Among University Students: A Prospective Cohort Study
Brief Title: Assocation Between In-person Instruction and COVID-19 Risk
Acronym: Campus&Corona
Status: Completed | Type: Observational
Sponsor: Oslo Metropolitan University (Other)
Collaborators: Norwegian Institute of Public Health (Other Government)
Responsible Party: Principal Investigator, Atle Fretheim, Adjunct Professor, Oslo Metropolitan University
Other Study IDs: 172155
Record Dates: First submitted 2020-08-25; First posted 2020-08-27 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Infection; Infection Control
Keywords: COVID-19; Social distancing; Digital instruction; In-person instruction; Campus; University; College; Higher education institutions
MeSH Terms: conditions — Infections; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (14):
- Students, Higher Education Institution 1: All first, second, and third year students at Higher Education Institution 1 who agree to take part in study.
  Interventions: Behavioral: Online instruction; Behavioral: In-person instruction
- Students, Higher Education Institution 2: All first, second, and third year students at Higher Education Institution 2 who agree to take part in study.
  Interventions: Behavioral: Online instruction; Behavioral: In-person instruction
- Students, Higher Education Institution 3: All first, second, and third year students at Higher Education Institution 3 who agree to take part in study.
  Interventions: Behavioral: Online instruction; Behavioral: In-person instruction
- Students, Higher Education Institution 4: All first, second, and third year students at Higher Education Institution 4 who agree to take part in study.
  Interventions: Behavioral: Online instruction; Behavioral: In-person instruction
- Students, Higher Education Institution 5: All first, second, and third year students atHigher Education Institution 5 who agree to take part in study.
  Interventions: Behavioral: Online instruction; Behavioral: In-person instruction
- Students, Higher Education Institution 6: All first, second, and third year students at Higher Education Institution 6 who agree to take part in study.
  Interventions: Behavioral: Online instruction; Behavioral: In-person instruction
- Students, Higher Education Institution 7: All first, second, and third year students at Higher Education Institution 7 who agree to take part in study.
  Interventions: Behavioral: Online instruction; Behavioral: In-person instruction
- Students, Higher Education Institution 8: All first, second, and third year students at Higher Education Institution 8 who agree to take part in study.
  Interventions: Behavioral: Online instruction; Behavioral: In-person instruction
- Students, Higher Education Institution 9: All first, second, and third year students at Higher Education Institution 9 who agree to take part in study.
  Interventions: Behavioral: Online instruction; Behavioral: In-person instruction
- Students, Higher Education Institution 10: All first, second, and third year students at Higher Education Institution 10 who agree to take part in study.
  Interventions: Behavioral: Online instruction; Behavioral: In-person instruction
- Students, Higher Education Institution 11: All first, second, and third year students at Higher Education Institution 11 who agree to take part in study.
  Interventions: Behavioral: Online instruction; Behavioral: In-person instruction
- Students, Higher Education Institution 12: All first, second, and third year students at Higher Education Institution 12 who agree to take part in study.
  Interventions: Behavioral: Online instruction; Behavioral: In-person instruction
- Students, Higher Education Institution 13: All first, second, and third year students at Higher Education Institution 13 who agree to take part in study.
  Interventions: Behavioral: Online instruction; Behavioral: In-person instruction
- Students, Higher Education Institution 14: All first, second, and third year students at Higer Education Institution 14 who agree to take part in the study.
  Interventions: Behavioral: Online instruction; Behavioral: In-person instruction

INTERVENTIONS:
Behavioral: Online instruction — For some courses and groups of students, instruction is primarily offered digitally, so that the students can participate from outside campus.
Behavioral: In-person instruction — For some courses and groups of students, instruction is primarily offered in-person, on campus (or elsewhere).

SUMMARY:
Whether university teaching on campus with infection control measures in place is associated with higher risk of COVID-19 than online instruction, is unknown. The investigators will assess this by conducting repeated surveys among students at universities and university colleges in Norway, where some instruction is given in-person, and some is provided online (hybrid model). The investigators will ask about the students' COVID-19 status, and how much in-person and online instruction the students are getting. The investigators will estimate the association between in-person instruction and COVID-19-risk using multivariate regression, controlling for likely confounders. The investigators will also assess whether type of instruction is associated with how satisfied the students are with the instruction the students are offered, their quality of life, and learning outcomes.

DETAILED DESCRIPTION:
The investigators are inviting all universities and university colleges in Norway to take part. All students at institutions that agree to participate will receive an SMS (alternatively an e-mail) inviting them to take part in the study. The invitation includes a link that directs participants to a web-based informed consent-form and questionnaire. The investigators will use the University of Oslo's solutions for online consent form, web-based survey (Nettskjema), and secure storage of research data (TSD).

The investigators will ask the participants if the participants have been tested for COVID-19, the results of such a test, how much in-person instruction the students have been offered, and how much online instruction the students have been offered. The investigators will also inquire about other risk factors for COVID-19 and background variables that may be included as potential adjustment factors (confounders) in the analyses (see Attachment 1 - Questionnaire).

The investigators will survey the students every two weeks by new invitations by SMS or e-mail. The study period will last as long as the universities maintain their arrangement with in-person instruction for only select groups of students. The investigators plan for a study period that lasts for the remainder of 2020. The investigators will ask for the participants consent to link the survey results to information on study programme, basis for admission, study status, academic results, sex and age from the Common Student System.

The investigators will run multivariate regressions to test whether there is an association between in-person instruction and the outcomes.

In-person instruction is a continuous variable, defined as

(Number of days offered in-person instruction) / (Number of days offered in-person instruction + Number of days offered online instruction)

The investigators will control for potentially confounding variables, including year of study program, field of study, age, and gender. The investigators plan for separate analyses for each participating university/university college, and a pooled analysis across institutions.

ELIGIBILITY:
Inclusion Criteria:

* Student in first, second, or third year at university or university college
* Agrees to participate (signed consent form)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All university of university college students who agree to participate.
Sampling Method: Non-Probability Sample
Enrollment: 26754 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
COVID-19 incidence | Through study completion, i.e. 4 months.
  Self-reported positive test results

SECONDARY OUTCOMES:
Quality of life | Through study completion, i.e. 4 months.
  Self-reported ("Overall, how satisfied are you with life right now?")
Satisfaction with teaching | Through study completion, i.e. 4 months.
  Self-reported ("Overall, how satisfied have you been with the teaching you have received in the past 14 days?")
COVID-19 testing incidence | Through study completion, i.e. 4 months.
  Self-reported
Learning outcome | End of term, December 2020.
  Exam results from Common Student System

CONTACTS AND LOCATIONS:
Overall Officials: Atle Fretheim, PhD, Principal Investigator — Oslo Metropolitan University
Locations (1):
- Oslo Metropolitan University, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
We plan to make the full data set publicly available, after ensuring the re-identification of individuals is not possible.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From spring 2021 and for at least 5 years.

REFERENCES:
- [Result] Fretheim A, Helleve A, Loyland B, Sandbekken IH, Flato M, Telle K, Watle SV, Schjoll A, Helseth S, Jamtvedt G, Hart RK. Relationship between teaching modality and COVID-19, well-being, and teaching satisfaction (campus & corona): A cohort study among students in higher education. Public Health Pract (Oxf). 2021 Nov;2:100187. doi: 10.1016/j.puhip.2021.100187. Epub 2021 Aug 27. PMID 34467258
- See also: Pre-print version of study report manuscript. — https://www.medrxiv.org/content/10.1101/2021.03.26.21254388v1